CLINICAL TRIAL: NCT03399188
Title: Fecal Microbiota Transplantation and Analysis of Fecal Microbiome in IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0223
Record Dates: First submitted 2017-12-18; First posted 2018-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases, Fecal microbiota transplantation, microbiome
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Inflammatory bowel disease patients in active stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT group (Experimental): Group who received fecal microbiome transplantation
  Interventions: Procedure: Fecal microbiome transplantation

INTERVENTIONS:
Procedure: Fecal microbiome transplantation — Fecal microbiota transplantation will be performed through colonoscopy to the IBD patients. Donor feces will be extensively screened for other diseases. Colonoscopy will be done at FMT center of Severance Children's Hospital twice with a month of duration. Recipients will be admitted the day before colonoscopy, and they will be discharged after a day of observation.

SUMMARY:
Fecal microbiome of donor and recipient will be analyzed before and after fecal microbiota transplantation in IBD patients.

DETAILED DESCRIPTION:
Fecal microbiota transplantation will be performed to the IBD patients, and microbial analysis will be done for donor and recipient feces. Fecal microbiota transplantation will be done twice via colonoscopy, with one month of duration. During the early stage of Fecal microbiota transplantation, recipient feces will be analyzed for the intestinal microbiota frequently.

Clinical outcome will be assessed 1month, 2month, 6month, and 1 year after the transplantation.

Relevance of intestinal microbial change and clinical outcome after transplantation and factors associated with successful clinical outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 7 years old to 80 years old at start of trial
* Inflammatory bowel disease such as ulcerative colitis, Crohn's disease, and Behcet's colitis
* Patients who do not respond to the conventional treatments or who do not wish/not able to use one.
* Patients who agree to participate in the trial after thorough explanation
* Evidence of active disease

Exclusion Criteria:

* Patients whose CRP<8, calprotectin<200, and mucosal healing endoscopically (who are in stable state)
* Patients whose symptom is due to other disease than IBD

  _Patients with immunosuppressive disease
* Patients who are clinically unstable such as massive hemorrhage or perforation
* Patients with toxic megacolon, paralytic ileus, or symptomatic intestinal obstruction
* Absolute neutrophil count (ANC) <1.5 *10^9/L (1500/mm3)
* Pregnant or under breast feeding
* Patients enrolled in other clinical trials

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 6months after the Second FMT
  For Ulcerative Colitis patients Patients 18 years old and under: Pediatric ulcerative colitis activity index (PUCAI) less than 10.
  It ranges from 0 to 85, with a higher score indicating greater severity of disease Patients over 18 years old: Partial Mayo score same or less than 1 It ranges from 0 to 9, with a higher score indicating greater severity of disease For Crohn's Disease patients Patients 18 years old and under: Pediatric Crohn's disease activity index (PCDAI) less than 10 It ranges from 0 to 100, with a higher score indicating greater severity of disease Patients over 18 years old: Crohn's disease activity index (CDAI) less than 150 It ranges from 0 to over 600, with a higher score indicating greater severity of disease

SECONDARY OUTCOMES:
Microbiome analysis by using relative abundance at phylum and genus level, beta diversity | Before, day 0~28 of 1st FMT, day 0~28, 60, 90, 180 of 2nd FMT
  * Microbial changes (increase of microbial diversity and improvement of firmicutes/bacteriodes ratio) in an early stage after FMT by using Relative abundance at phylum and genus level
  * Microbial stability after FMT for one week (change in beta diversity)
Clinical response using disease activity index | 6 months after the Second FMT
Endoscopic healing | 4 weeks after the First FMT
Adverse events | 6 months after the Second FMT
  Any adverse events thought to be related to FMT will be measured throughout the follow-up period after FMT.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided